CLINICAL TRIAL: NCT06475222
Title: Development and Effectiveness Evaluation of Facial Serum and Mask and Ready-to-drink Jelly From Thai Rice (Oryza Sativa L.)
Brief Title: Facial Serum and Mask and Ready-to-drink Jelly From Thai Rice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burapha University (Other)
Responsible Party: Principal Investigator, Piyapong Prasertsri, Associate Professor Dr., Burapha University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IRB1-047/2567
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Rice Serum; Rice Mask; Rice Jelly
Keywords: Thai rice

STUDY DESIGN:
Intervention Model Description: Study 1 is single group model, study 2 is parallel model, and study 3 is crossover model.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Study 1: Facial serum with alpha albutin (Active Comparator): Participants will be randomly applied with home-based program of facial serum producing from 2% alpha albutin (standard facial serum) on either right side or left side of their face daily for 12 weeks.
  Interventions: Other: Study 1: Facial serum with alpha albutin
- Study 1: Facial serum with Tubtim Chumpae rice extract (Experimental): Participants will be randomly applied with home-based program of facial serum producing from Tubtim Chumpae rice extract on either right side or left side of their face daily for 12 weeks.
  Interventions: Other: Study 1: Facial serum with Tubtim Chumpae rice extract
- Study 2: Facial mask with Hom Pathum rice extract (Experimental): Participants will receive home-based program of facial mask with Hom Pathum rice extract for 30 min/day, 2 days/week for 12 weeks.
  Interventions: Other: Study 2: Facial mask with Hom Pathum rice extract
- Study 3: Control jelly (Active Comparator): Participants will consume with control jelly at 3.5 g/kg body weight. Consumption will be taken at Burapha University.
  Interventions: Other: Study 3: Control jelly
- Study 3: Jelly with Tubtim Chumpae rice (Experimental): Participants will consume with Tubtim Chumpae rice jelly at 3.5 g/kg body weight. Consumption will be taken at Burapha University.
  Interventions: Other: Study 3: Jelly with Tubtim Chumpae rice
- Study 3: Jelly with Hom Pathum rice (Experimental): Participants will consume with Hom Pathum rice jelly at 3.5 g/kg body weight. Consumption will be taken at Burapha University.
  Interventions: Other: Study 3: Jelly with Hom Pathum rice

INTERVENTIONS:
Other: Study 1: Facial serum with alpha albutin — Applying with facial serum with 2% alpha albutin as active comparator daily for 12 weeks.
  Arms: Study 1: Facial serum with alpha albutin
Other: Study 1: Facial serum with Tubtim Chumpae rice extract — Applying with facial serum with Tubtim Chumpae rice extract as experimental intervention daily for 12 weeks.
  Arms: Study 1: Facial serum with Tubtim Chumpae rice extract
Other: Study 2: Facial mask with Hom Pathum rice extract — Applying with facial mask with Hom Pathum rice extract as experimental intervention for 30 min/day, 2 days/week for 12 weeks.
  Arms: Study 2: Facial mask with Hom Pathum rice extract
Other: Study 3: Control jelly — Consumption with control jelly as active comparator at 3.5 g/kg body weight.
  Arms: Study 3: Control jelly
Other: Study 3: Jelly with Tubtim Chumpae rice — Consumption with jelly with Tubtim Chumpae rice as experimental intervention at 3.5 g/kg body weight.
  Arms: Study 3: Jelly with Tubtim Chumpae rice
Other: Study 3: Jelly with Hom Pathum rice — Consumption with jelly with Hom Pathum rice as experimental intervention at 3.5 g/kg body weight.
  Arms: Study 3: Jelly with Hom Pathum rice

SUMMARY:
This study consisted of three sub-studies including 1) development and evaluation of facial serum from Thai rice on skin moisture, elasticity, oiliness, and melanin in healthy participants 2) development and evaluation of facial mask from Thai rice on skin moisture, elasticity, oiliness, and melanin in healthy participants and 3) development and evaluation of ready-to-drink jelly from Thai rice on controlling blood glucose and endurance time in healthy participants.

DETAILED DESCRIPTION:
Study 1: 30 male and female participants, age 30-50 years will be randomly applied with facial serum producing from either 2% alpha albutin (standard facial serum) or Tubtim Chumphae rice extract on either right side or left side of their face daily for 12 weeks.

Study 2: 60 male and female participants, age 30-50 years will be randomly assigned into 2 groups including 1) control group (n = 30): participants will not receive any facial mask for 12 weeks and 2) treatment group (n = 30): participants will be applied with home-based program facial mask with Hom Pathum rice extract for 30 min/day, 2 days/week for 12 weeks.

Study 3: this study consists of 2 sub-studies. Study 3.1: 25 male and female participants, age 18-35 years will be randomly consumed with control jelly, jelly with Tubtim Chumphae rice, and jelly with Hom Pathum rice at 3.5 g/kg body weight. All participants will be measured for blood glucose levels before consumption and after consumption at 30, 60, 90, and 120 min. Study 3.2: 25 male and female participants, age 18-35 years will be randomly consumed with control jelly, jelly with Tubtim Chumphae rice, and jelly with Hom Pathum rice at 3.5 g/kg body weight. After each consumption, all participants will perform walking or running on treadmill at intensity of 80% maximal heart rate to measure maximal oxygen consumption.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age between 18 to 50 years
* Healthy
* Interested in facial serum with Thai rice extract or facial mask with Thai rice extract or jelly from with Thai rice

Exclusion Criteria:

* History of adverse effects from facial serum or mask application or jelly consumption
* Skin allergy
* Skin disorders
* Skin wounds
* History of allergy to Thai rice, particularly in Tubtim Chumpae and Hom Pathum
* History of allergy to facial serum or mask, i.e., serum or mask from rice
* History of allergy to gelatin
* Signs or symptoms of fever or infection
* Abnormal body mass index
* Regular smokers or alcohol drinkers (>2 times per week)
* Regular exerciser (>2 times per week or >150 min per week)
* Regular intake of dietary supplements, i.e., vitamins, antioxidants
* Hypertension, diabetes, cardiovascular disease, respiratory disease, endocrine disease, neuromuscular disease, musculoskeletal disease, liver disease, renal disease, immune disease, infectious disease, or cancer

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Level of skin moisture | Before intervention, immediately after intervention, ends of week 4, week 8, and week 12]
  Studies 1 and 2 determine level of skin moisture in arbitrary unit (no unit) using Multiprobe Adapter System with Corneometer® CM 825 probe.
Level of skin elasticity | Before intervention, immediately after intervention, ends of week 4, week 8, and week 12]
  Studies 1 and 2 determine level of skin elasticity in arbitrary unit (no unit) using Multiprobe Adapter System with Cutometer® 580 probe.
Level of skin oiliness | Before intervention, immediately after intervention, ends of week 4, week 8, and week 12]
  Studies 1 and 2 determine level of skin oiliness in arbitrary unit (no unit) using Multiprobe Adapter System with Sebumeter® SM 815 probe.
Level of skin melanin | Before intervention, immediately after intervention, ends of week 4, week 8, and week 12]
  Studies 1 and 2 determine level of skin melanin in arbitrary unit (no unit) using Multiprobe Adapter System with Mexameter® MX18 probe.
Level of blood glucose | Before jelly consumption and after jelly consumption at 30, 60, 90, and 120 minutes
  Study 3.1 determines level of blood glucose in mg/dL unit
Level of maximal oxygen consumption | After jelly consumption for 30 minutes
  Study 3.2 determines level of maximal oxygen consumption in mL/kg/min unit by walking or running on treadmill at intensity of 80% maximal heart rate.
Concentration of interferon-gamma | Before and immediately after maximal oxygen consumption test
  Study 3.2 determines concentration of interferon-gamma in serum in pg (picogram)/mL unit
Concentration of tumor necrosis factor-alpha | Before and immediately after maximal oxygen consumption test
  Study 3.2 determines concentration of tumor necrosis factor-alpha in serum in pg (picogram)/mL unit
Concentration of interleukin-10 | Before and immediately after maximal oxygen consumption test
  Study 3.2 determines concentration of interleukin-10 in serum in pg (picogram)/mL unit
Level of superoxide dismutase activity | Before and immediately after maximal oxygen consumption test
  Study 3.2 determines level of superoxide dismutase activity in percentage (%) unit
Concentration of malondialdehyde | Before and immediately after maximal oxygen consumption test
  Study 3.2 determines concentration of malondialdehyde in micromolar (uM) unit

CONTACTS AND LOCATIONS:
Overall Officials: Piyapong Prasertsri, Ph.D., Principal Investigator — Burapha University
Locations (1):
- Piyapong Prasertsri, Mueang, Changwat Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.